CLINICAL TRIAL: NCT04319640
Title: the Effects of Sleep Intervention in Children With Autism Spectrum Disorder Through Synchronized Eye-tracking and Functional Near-infrared Spectroscopy
Brief Title: Cognitive Behaviour Therapy for Sleep Problems in Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Sijia Gu, staff of Research Department, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCMCIRB-K2018040
Record Dates: First submitted 2020-02-06; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder; Cognitive Behaviour Therapy
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: 1:1 parallel randomized controlled trial
Who Masked: Participant
Masking Description: Participant blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBTI (Experimental): N= 80 participants are offered Cognitive behaviour therapy for insomnia (CBT-I)
  Interventions: Behavioral: Cognitive behaviour therapy for insomnia; Behavioral: psychoeducation for ASD
- psychoeducation (Active Comparator): N= 80 participants are offered psychoeducation about information on ASD
  Interventions: Behavioral: psychoeducation for ASD

INTERVENTIONS:
Behavioral: Cognitive behaviour therapy for insomnia — CBT-I for children with ASD includes sleep hygiene, restriction of time in bed, stimulus control, cognitive therapy, and relaxation techniques. The treatment consists of 5 weekly modules.
  Arms: CBTI
Behavioral: psychoeducation for ASD — psychoeducation contains information about ASD, The treatment consists of 5 weekly modules.

SUMMARY:
Sleep disturbance is very common in children with autism spectrum disorder (ASD),and closely associated with their core symptom, social deficit.This trial investigates the effects of Cognitive behaviour therapy for insomnia (CBT-I) in children with autism spectrum disorder with sleep problems through synchronized eye-tracking and functional near-infrared spectroscopy (fNIRS). This is a 1:1 parallel single-blind randomized controlled trial.

DETAILED DESCRIPTION:
sleep disturbance is significantly associated with social deficit of ASD and but the congnitive-neural mechanism underlying this association remains unclear. Cognitive behaviour therapy for insomnia (iCBT-I) is considered as an evidence-based treatment for insomnia. After 5 consecutive sleep interventions is a 2-year following up study, the above issue is further tested with emphasis on progressive trajectory from a developmental perspective. we examine the influence of sleep disturbance on face processing and neural response during naturalistic social behavior of ASD children using synchronized eye-tracking and functional near-infrared spectroscopy (fNIRS) to uncover the neural mechanism for that sleep disturbance influences social deficit.

ELIGIBILITY:
Inclusion Criteria:

1. meet the diagnostic criteria for autism DSM-5 and ADOS-2;
2. age 24months to 59months s old;
3. willing to participate in this study, and can complete the following assessments at the specific time.

Exclusion Criteria:

Exclusion of severe respiratory diseases, schizophrenia, epilepsy and other brain diseases;

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
congnitive-neural outcomes | changes from baseline, 6 months after the intervention, 12 months after the intervention and 6 year olds
  The investigators examine the influence of sleep disorders on face processing and neural response at baseline, 6 months after the intervention, 12 months after the intervention and when children 6 year olds by synchronized eye-tracking and functional near-infrared spectroscopy (fNIRS) to uncover the neural mechanism for that sleep disturbance influences social-emotional development.
ADOS-2 | changes from baseline, 6 months after the intervention, 12 months after the intervention and 6 year olds
  The ADOS-2 is the standard instrument for assessing autism spectrum disorders (ASD) across age, developmental level, and language skills.

SECONDARY OUTCOMES:
Sleep diaries by using Actigraphy | changes from baseline, 6 months after the intervention, 12 months after the intervention and 6 year olds
  Different sleep parameters, such as sleep onset latency (SOL) and wake after sleep onset (WASO) will be determined using wrist actigraphy. Participants will be provided with an actiwatch at baseline, 6 months after the intervention , 12 months after the intervention and when children 6 year olds . The actiwatch will be worn on the non-dominant arm 24 hours a day, except for while bathing, during the 1-week screening periodmovement and nighttime sleep parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Jiang, PhD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- shanghai children's medicial center affiliated shanghai jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China